CLINICAL TRIAL: NCT07078617
Title: Comparison of PNF and Soft Tissue Mobilization Techniques Along With Exercise for the Treatment of Bell's Palsy
Brief Title: Effectiveness of PNF and STM in Bell Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elite College of Management Sciences, Gujranwala, Pakistan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-GCUF-079348
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Bell's Palsy
Keywords: Facial disability index; PNF; House Brackmann scale
MeSH Terms: interventions — Muscle Stretching Exercises; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation (Experimental): Repeated stretch and Hold relax method used in this technique.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation
- Soft Tissue Mobilization along with exercise (Experimental): Effleurage, Kneading and hacking along with facial exercises
  Interventions: Other: Soft Tissue Mobilization along with exercise

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation — PNF technique given for 3-4 days/week and electrical stimulation of DL-2 stimulator with 90 repetitions on each motor point of facial muscle for 3-4 days/week.
  Arms: Proprioceptive Neuromuscular Facilitation
Other: Soft Tissue Mobilization along with exercise — Soft tissue mobilization along with facial exercise 3- days/ week and electrical stimulation of DL-2 stimulator with 90 repetitions on each motor point of facial muscle for 3-4 days/week.
  Arms: Soft Tissue Mobilization along with exercise

SUMMARY:
Our study aims to determine the efficacy of PNF and Soft tissue mobilization techniques with exercise for Bell's palsy. It ascertains which intervention yields better outcomes and has greater effect on recovery.

DETAILED DESCRIPTION:
It is a randomized controlled trial. This study includes 28 participants allocated into two groups by coin tossing method. Group A receives PNF and Group B receives soft tissue mobilization along with exercise. Both of the groups receive electrical stimulation as baseline treatment. The assessment of participants is done by using facial disability index and House Brackmann scale.

ELIGIBILITY:
Inclusion Criteria:

* aged 25-50 years
* sudden onset of one-sided Bell's palsy
* Ability and Eagerness to provide informed consent in written form

Exclusion Criteria:

* Uncontrolled Hypertension
* Uncooperative patients and those who don't follow instructions.
* Previous mental disorder that may affect participation.
* Preexisting ear surgery

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Facial disability index | 4 weeks
  in 1996, this scale was invented. This tool is used to evaluate functional and psychological effects of cranial nerve VII dysfunction like Bell's palsy. It consists of two subscales one is Physical Function and second is Social/Wellbeing Function, each with a range 0 to 100 where higher score shows better function and lesser disability.

SECONDARY OUTCOMES:
House Brackmann scale | 4 weeks
  This scale was invented in 1985 by DE Brackmann and Dr.John W.House. This scale is used to evaluate the severity of cranial nerve VII. it consists of six grades. Grade 1 indicates Normal and Grade 6 indicates complete paralysis.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Rafiq, PhD, Principal Investigator — Elite College of Management sciences
Locations (1):
- Al Raee Hospital Gujranwala, Salamat Hospital Gujranwala, Chaudhary Hospital Gujranwala, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amjad A, Jamil A, Fatima N, Javaid HB, Zahid H. Effects of Kabat rehabilitation versus mime therapy on facial disability and synkinesis in patients of Bell's palsy. J Pak Med Assoc. 2024 Nov;74(11):1927-1931. doi: 10.47391/JPMA.11247. PMID 39548608
- [Result] Burelo-Peregrino EG, Salas-Magana M, Arias-Vazquez PI, Tovilla-Zarate CA, Bermudez-Ocana DY, Lopez-Narvaez ML, Guzman-Priego CG, Gonzalez-Castro TB, Juarez-Rojop IE. Efficacy of electrotherapy in Bell's palsy treatment: A systematic review. J Back Musculoskelet Rehabil. 2020;33(5):865-874. doi: 10.3233/BMR-171031. PMID 32144972
- [Result] Khan AJ, Szczepura A, Palmer S, Bark C, Neville C, Thomson D, Martin H, Nduka C. Physical therapy for facial nerve paralysis (Bell's palsy): An updated and extended systematic review of the evidence for facial exercise therapy. Clin Rehabil. 2022 Nov;36(11):1424-1449. doi: 10.1177/02692155221110727. Epub 2022 Jul 5. PMID 35787015
- [Result] Albishi AM, Altowairqi RT, Alhadlaq SA, Alsulboud SK, Alhusaini AA, Alokaily AO, Alotibi M. Cross-cultural adaptation, reliability, and validation of the Arabic version of the Motor Activity Log (MAL-30) Scale in patients with stroke in Saudi Arabia. Disabil Rehabil. 2025 Dec;47(26):7042-7050. doi: 10.1080/09638288.2025.2526701. Epub 2025 Jul 3. PMID 40607587
- [Result] Eviston TJ, Croxson GR, Kennedy PG, Hadlock T, Krishnan AV. Bell's palsy: aetiology, clinical features and multidisciplinary care. J Neurol Neurosurg Psychiatry. 2015 Dec;86(12):1356-61. doi: 10.1136/jnnp-2014-309563. Epub 2015 Apr 9. PMID 25857657